CLINICAL TRIAL: NCT02913456
Title: A European Disease Registry Study to Prospectively Observe Treatment Patterns and Outcomes in Patients With HER2-Positive Unresectable Locally Advanced or Metastatic Breast Cancer
Brief Title: A European Registry Study to Prospectively Observe Treatment Patterns and Outcomes in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Unresectable Locally Advanced (LA) or Metastatic Breast Cancer (mBC) (SAMANTHA)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: MO39146
Record Dates: First submitted 2016-09-22; First posted 2016-09-23 (Estimated); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- HER2-positive unresectable LA/mBC: Participants with HER2-positive unresectable LA/mBC diagnosed up to 6 months prior to enrollment will be included in the study. Enrolled participants will receive treatment and clinical assessments for their HER2-positive unresectable LA/mBC as determined by their treating physician, according to the standard of care and routine clinical practice at each site.

SUMMARY:
This disease registry is a prospective, multicenter non-interventional study designed to observe anti-cancer treatment regimens and clinical outcomes in participants with HER2-positive unresectable LA/mBC. Diagnosis of unresectable LA or mBC can be up to 6 months old prior to registry enrollment.

ELIGIBILITY:
Inclusion Criteria:

- Initially diagnosed with HER2-positive unresectable LA/mBC no more than 6 months prior to enrollment, although they can have received anti-cancer treatment during that time

Exclusion Criteria:

- Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants initially diagnosed with HER2-positive unresectable LA/mBC no more than 6 months prior to enrollment
Sampling Method: Non-Probability Sample
Enrollment: 629 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival per Anti-cancer Treatment Regimens Assessed According to Site-/Country-Specific Medical Practice | Baseline up to 8 years
Percentage of Participants by Different Anti-cancer Treatment Regimens and Treatment Sequences | Baseline up to 8 years

SECONDARY OUTCOMES:
Overall Survival | Baseline up to 8 years
Duration of Response per Anti-cancer Treatment Regimens Assessed According to Site-/Country-Specific Medical Practice | Baseline up to 8 years
Percentage of Participants with Best Overall Response of Complete Response (CR) or Partial Response (PR) per Anti-cancer Treatment Regimens Assessed According to Site-/Country-Specific Medical Practice | Baseline up to 8 years
Total Number of Treatment Regimens Received by Participants | Baseline up to 8 years
Percentage of Participants with Adverse Events (AEs), Serious AEs, and Protocol-defined AEs of Special Interest | Baseline up to 8 years
Percentage of Participants with HER2 Re-testing of Metastases | Baseline up to 8 years
Percentage of Participants with Change in HER2 Status | Baseline up to 8 years
Percentage of Participants by Type of HER2 Testing (Immunohistochemistry and/or Fluorescence In situ Hybridization [FISH]) | Baseline up to 8 years
Percentage of Participants with Different Anti-Cancer Treatment Regimens by Country | Baseline up to 8 years
Percentage of Participants with History of Breast Cancer by Different Anti-Cancer Treatment Regimens | Baseline up to 8 years
EuroQol 5-Dimensions Questionnaire (EQ-5D) Score | Baseline up to 8 years
Functional Assessment of Cancer Therapy-Breast (FACT-B) Questionnaire Score | Baseline up to 8 years
Total Healthcare Cost | Baseline up to 8 years
Cost of Treating Associated AEs | Baseline up to 8 years
Resource Utilization: Percentage of Participants with Breast Cancer Associated Procedures | Baseline up to 8 years
Resource Utilization: Percentage of Participants with Hospitalization | Baseline up to 8 years
Resource Utilization: Percentage of Participants with Emergency Room Attendances and Outpatient Visits | Baseline up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (54):
- Austria (11):
  - Lkh-Univ. Klinikum Graz; Klinik Für Gynäkologie, Graz
  - LKH-UNIV. KLINIKUM GRAZ; Klinische Abteilung für Onkologie, Graz
  - Klinikum Klagenfurt; Abt. f. Hämatologie u. internistische Onkologie, Klagenfurt
  - LKH Hochsteiermark; Abt. für Hämato-Onkologie, Leoben
  - Ordensklinikum Linz Elisabethinen ; I. INTERNE ABT., Linz
  - A.Ö. Krankenhaus Der Barmherzigen Schwestern Ried; Interne Abtl., Ried-innkreis
  - Medizinische Universität Wien; Univ.Klinik für Frauenheilkunde - Klinik für Gynäkologie, Vienna
  - Medizinische Universität Wien; Univ.Klinik für Innere Medizin I, Vienna
  - Hanusch-Krankenhaus; Geburtshilfliche und Gynäkologische Abteilung, Vienna
  - A.Ö. Lhk Villach; Abt. Für Gynäkologie, Villach
  - Landesklinikum Wiener Neustadt; Innere Medizin, Hämatologie u. internistische Onkologie, Wiener Neustadt
- Bulgaria (11):
  - Multiprofile Hospital for Active Treatment Central Onco Hospital OOD, Plovdiv
  - Complex Oncological Center - Plovdiv, EOOD, Plovdiv
  - Mdozs - Russe, Rousse
  - MHAT Nadezhda, Sofia
  - Tokuda Hospital; Medical Oncology Department, Sofia
  - University Multiprofile Hospital for Active Treatment Tsaritsa Yoanna - ISUL EAD, Sofia
  - SHATOD - Sofia, Sofia
  - Complex Oncology Center-Burgas; Medical Oncology, Sofia
  - District Oncology Dispensary; Dept of Chimiotherapy, Stara Zagora
  - District Oncology Dispensary Wit Stationary, Varna
  - Comprehensive Oncology Center - Vratsa, Vratsa
- Italy (19):
  - Irccs Ist. Tumori Giovanni Paolo Ii; Dipartimento Oncologia Medica, Bari, Apulia
  - Ospedale Barletta - Mons. Dimiccoli; Dip. Oncologia, Barletta, Apulia
  - A.O. Universitaria Policlinico Di Modena; Oncologia, Modena, Emilia-Romagna
  - RCCS - Centro di Riferimento; Oncologia Medica B, Aviano (PN), Friuli Venezia Giulia
  - Ospedale S. Maria Goretti; Divisione Di Oncologia Medica, Latina, Lazio
  - Ospedale S.S. Trinità Nuovo; Divisione Oncologia, Sora, Lazio
  - Ospedale Belcolle Di Viterbo; Oncologia, Viterbo, Lazio
  - Az. Osp. Spedali Civili; Divisione Di Oncologia - Iii Medicina, Brescia, Lombardy
  - Ospedale Degli Infermi Di Biella; Reparto Oncologia Medica, Ponderano (BI), Piedmont
  - Ospedale Cannizzaro, Oncologia, Catania, Sicily
  - Casa Di Cura Di Alta Specialita La Maddalena; Dept. Oncologico Di Iii Livello, Palermo, Sicily
  - A.O.U. Ospedali Riuniti Umberto I-G.M.Lancisi-G.Salesi Ancona;S.O.D. MED.Interna-Clinica Oncologica, Ancona, The Marches
  - Azienda Ospedaliero-Universitaria Careggi; SOD Radioterapia, Florence, Tuscany
  - Ospedale San Luca; Oncologia, Lucca, Tuscany
  - Azienda Ospedaliera Di Perugia Ospedale s. Maria Della Misericordia; Oncologia Medica, Sant'Andrea Delle Fratte (PG), Umbria
  - Ospedale Civile; Oncologia Medica, Camposampiero, Veneto
  - Azienda Ospedaliero Universitaria di Ferrara - U.O. Di Oncologia, Cona (FE), Veneto
  - Azienda ULSS 21 Ospedale Mater Salutis; Dip. di Oncologia, Legnago (VR), Veneto
  - A.O.U. Integrata Verona - Policlinico G.B. Rossi; Oncologia Medica - Dip. di Medicina, Verona, Veneto
- Portugal (6):
  - Hospital Garcia de Orta; Servico de Oncologia Medica, Almada
  - IPO de Coimbra; Servico de Oncologia Medica, Coimbra
  - Hospital Santo Antonio dos Capuchos;Servico de Oncologia Medica, Lisbon
  - Hospital de Santa Maria; Servico de Oncologia Medica, Lisbon
  - Hospital Beatriz Angelo; Departamento de Oncologia, Loures
  - IPO do Porto; Servico de Oncologia Medica, Porto
- Romania (7):
  - County Hospital Alba; Oncology, Alba Iulia
  - "Filantropia" Clinical Hospital; Gynecological Oncology, Bucharest
  - Institutul Oncologic Prof. Dr. Al. Trestioreanu Bucuresti, Bucharest
  - Cluj-Napoca Emergency Clinical County Hospital; Medical Oncology, Cluj-Napoca
  - Prof. Dr. I. Chiricuta Institute of Oncology, Cluj-Napoca
  - Centrul de Oncologie Sfantul Nectarie, Craiova
  - Oncomed SRL, Timișoara